CLINICAL TRIAL: NCT03906279
Title: Automatic Measurements of Choroidal Thickness Change in Response to Physiological and Refractive Changes
Brief Title: Choroidal Thickness Change in Response to Physiological and Refractive Changes
Status: Active, not recruiting | Type: Observational
Sponsor: Wrocław University of Science and Technology (Other)
Collaborators: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ST002.2018
Record Dates: First submitted 2019-04-03; First posted 2019-04-08 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Refractive Errors; Accommodation Disorder
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Myopic participants
- Emmetropic participants
- Hyperopic participants

SUMMARY:
There is a great need for precise and repeatable measurements of the choroidal thickness. Including the diurnal physiological changes, accommodation and refractive error impact on those measurements.

ELIGIBILITY:
Inclusion Criteria:

* participants with refractive error
* willing and able to understand and sign an informed consent form

Exclusion Criteria:

* patient unable to participate in the study
* any disease that causes visual opacity of optic media that unable to perform OCT scanning
* current enrolment in another clinical trial/research project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with refractive error
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Submacular choroidal thickness | 1 day
  OCT EDI recorded scans will be proceed with the custom-made software to determine choroidal thickness in the submacular region.
Peripapillar choroidal thickness | 1 day
  OCT EDI recorded scans will be proceed with the custom-made software to determine choroidal thickness in the peripapillar region.

SECONDARY OUTCOMES:
Axial length of the globe | 1 day
  Measured with optical biometer (Lenstar)
Anterior chamber depth - optical biometry | 1 day
  Measured with optical biometer (Lenstar)
Phakic lens thickness | 1 day
  Measured with optical biometer (Lenstar)
White to white diameter | 1 day
  Measured with optical biometer (Lenstar)
Angle to angle diameter of anterior chamber | 1 day
  Measured with optical coherent tomography for anterior chamber
Anterior chamber depth - OCT | 1 day
  Measured with optical coherent tomography for anterior chamber
Corneal keratometry (steep meridian and its axis and flat meridian with its axis) | 1 day
  Keratometry from autorefractokeratometer, topography or tomography recordings, radius measured in mm, magnitude of corneal astigmatism measured in local changes of dioptric power.
Spherical ametropia with cylindrical power of correcting lenses | 1 day
  Subjective refraction made by trained optometrist. Spherical ametropia measured by dioptric power of spherical equivalent lens and magnitude of astigmatism measured in cylindrical dioptries of correcting lens with its axis. Mode of notation: sphero-cylinder with negative cylinder (e.g. +0.50DS -0.50DC 180ax)
Best-corrected visual acuity | 1 day
  examined on ETDRS charts different for right and left eye

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Przeździecka-Dołyk, PhD, Principal Investigator — Wrocław University of Science and Technology
Locations (1):
- Department of Optics and Photonics, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
We intend to share anonymised data